CLINICAL TRIAL: NCT07247851
Title: Title of the Protocol: Combined Use of Vaginal Clindamycin Cream and Oral Metronidazole Versus Oral Metronidazole in Treatment of Bacterial Vagionosis: A Randomized Controlled Clinical Trial
Brief Title: Title of the Protocol: Combined Use of Vaginal Clindamycin Cream and Oral Metronidazole Versus Oral Metronidazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Gamal Anwar Elskaan, Lecturer of Obstetrics and Gynecology at Faculty of Medicine, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bacterial Vagionos
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-01

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — clindamycin phosphate; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Clindamycine with Metronidazole) (Active Comparator): About 50 female patients used Vaginal Clindamycin vaginal cream: 2% and Oral Metronidazole tablets in the treatment of Bacterial Vaginosis
  Interventions: Drug: Clindamycin Phosphate
- Group B (Metronidazole) (Active Comparator): About 50 female patients used Metronidazole tables in the treatment of Bacterial Vaginosis
  Interventions: Drug: Clindamycin Phosphate

INTERVENTIONS:
Drug: Clindamycin Phosphate — comparing the efficacy of the combined use of vaginal clindamycin cream and oral metronidazole in comparison to oral metronidazole alone for bacterial vaginosis treatment.
  Other Names: Metronidazole

SUMMARY:
Bacterial vaginosis (BV) constitutes a gynecological condition characterized by an alteration of the vaginal microenvironment and more specifically an alteration of the normal Lactobacillus-dominated vaginal flora, to a flora that includes a variety of facultative and obligatory anaerobic bacteria; this alteration causes offensive smelling vaginal discharge, leading to significant psychological distress and a reduction in quality of life and may be associated with adverse outcomes following a gynecological/obstetrical surgical intervention, such as an increased risk of post-operative infections after pelvic surgery.

It has been observed in 29% of reproductive-age individuals in the United States, and the prevalence of BV varies with race and ethnicity

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) constitutes a gynecological condition characterized by an alteration of the vaginal microenvironment and more specifically an alteration of the normal Lactobacillus-dominated vaginal flora, to a flora that includes a variety of facultative and obligatory anaerobic bacteria

symptoms in cases of symptomatic BV include an elevated vaginal pH, grey-white milky vaginal discharge, itching, and a "fishy" odor. moreover, It is well known that unfavorable outcomes of early pregnancy including premature rupture of membranes (PROM), chorioamnionitis, preterm delivery, spontaneous abortion, and low birth weight can be exacerbated by BV during pregnancy.

Aside from the evaluation of clinical symptoms, the gold standard for the confirmation of BV diagnosis is the Nugent score based on Gram staining and observing the number of lactobacilli and other morphotypes (different shapes of gardenerellavaginalis, prevotella species, and mobiluncus) which are scored between 0 and 10, where scores 7-10 show BV. However, traditional assessment using Nugent scoring typically requires more time, resources, and expertise, which can impact its use in a clinical setting. The preferred alternative in practice is the Amsel scoring or a Gram stain.

The Amsel scoring system is simple to use and is based on four predefined criteria: (I) the presence of homogeneous, thin, greyish white vaginal discharge, (II) a vaginal pH over 4.5, (III) a positive whiff-amine test, and (IV) >20% clue cells/high power field on a wet mount of vaginal secretions. Yet, important diagnostic tools for BV are the phase contrast microscope and a trained user.

Oral divided dose metronidazole is the most widely used therapy and serves as the standard of care for bacterial vaginosis. Despite its favorable pharmacodynamics, recurrence rates of BV are high, 69-80% within 12 months. The causes of recurrence are still not known, whether from development of a treatment resistant bacterial biofilm on the vaginal mucosa, reinfection from a sexual partner, or host factors leading to failure to re-establish the normal vaginal flora.Two-thirds of cases complain from bacterial vaginosis recurrence within a year of treatment.

Metronidazole treatment is also associated with side effects which can limit acceptability and adherence. Patients also dislike taking multiple courses of antibiotics and are concerned that they may acquire resistant bacteria. Preventing and reducing antimicrobial resistance is also a public health priority through improving antibiotic stewardship including a reduction in antibiotic use. The limited efficacy of current treatment for bacterial vaginosis and a need to reduce antibiotic exposure highlight the need for alternative therapies.

Clindamycin phosphate was approved by the united states (U.S) Food and Drug Administration (FDA) in 2021 for the treatment of bacterial vaginosis. It is unique among bacterial vaginosis treatments in that it is a thermosetting bioadhesive intravaginal cream formulated with 2% clindamycin phosphate designed to release the active ingredient for an extended period of time. Reduced leakage should result in better user compliance, and, because clindamycin is more effective with increased exposure time, the increased retention time is supposed to result in higher cure rates

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years with a clinical diagnosis and laboratory diagnosis as (cervical smear & high vaginal swab) of bacterial vaginosis.
* Diagnosed with Bacterial vaginosis the Amsel scoring system which requires 3 criteria of 4 criteria for diagnosis.:
* The presence of homogeneous, thin, greyish white vaginal discharge.
* Vaginal pH over 4.5.
* Positive whiff-amine test (the presence of a fishy odor following addition of KOH to the vaginal sample).
* More than 20% clue cells/high power field on a wet mount of vaginal secretions.

Exclusion Criteria:

* Other types of infections based on history and clinical examination as candida vaginitis (itching with cottage cheese whitish discharge, Trichomonas vaginalis (with yellowish green offensive discharge) and any sexually transmitted disease (STDs) as gonorrhea(watery creamy greenish discharge, pain on micturation)syphilis(appearance of shung-kur ulcer, painless sore), chlamydia(abnormal discharge from vagina, burning sensation on peeing, abnormal discharge from penis) or genital herpes (tingling, burning, itching around genitals on both parteners).
* Pregnant and lactating females
* Any contraindication or hypersensitivity to metronidazole use
* Use of other antibiotics or systemic antifungal agents within the previous 2 weeks or planned use within 2 weeks
* Use of topical vaginal antibiotics, antifungals or acidifying products recently or planned within 2 weeks
* Atrophic vaginitis
* Using IUD as contraceptive method because IUD is a risk factor for infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Bacterial Vaginosis treatment | At 2 weeks and through 6 months
  Assessment of the female patients whom suffering from Bacterial Vaginosis by Complete history description to changes of discharge odour and symptoms of vulvovaginitis as itching. and efficacy of both medications (reliving symptoms of BV as discharge & odour) .

CONTACTS AND LOCATIONS:
Overall Officials: Laila Aly Farid, Professor, Study Chair — Obstetrics and Gynecology, Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided